CLINICAL TRIAL: NCT05985720
Title: Evaluation of Cardiac Biomarkers and the Left and Right Ventricular Systolic and Diastolic Function in Asthmatic Children in Assuit University Hospital
Brief Title: Evaluation of Cardiac Biomarkers and Ventricular Function in Asthmatic Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Khalaf Saber, Principal Investigator, Assiut University
Other Study IDs: Asthmatic children
Record Dates: First submitted 2023-03-30; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Ventricular Dysfunction; Asthma in Children
Keywords: asthma; cardiac affection
MeSH Terms: conditions — Ventricular Dysfunction; Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation of cardiac biomarkers and the left and right ventricular systolic and diastolic function in asthmatic children in Assuit university hospital

DETAILED DESCRIPTION:
Severe acute asthma which is defined asthma that is uncontrolled despite maximal optimized therapy and treatment of contributory factors, or that worsens when high dose treatment is decreased(1) and it is characterized by severe respiratory distress because of increasing bronchoconstriction, leading to ventilation perfusion mismatch, hypoxia, respiratory muscle fatigue, carbon dioxide retention and respiratory acidosis(2) In acute severe asthma, the use of beta 2 agonists, together with hypoxia and tachycardia might cause increased myocardial workload further leading to myocardial infarction(3).

Cardiac biomarkers including Brain Natriuretic Peptide (BNP),Troponin I (TnI) and Creatine kinase muscle/brain(CK-MB) are used to detect myocardial injury(4).

The objective of the present study was to find out the incidence of myocardial dysfunction in patients of acute severe bronchial asthma based on cardiac biomarker levels at admission and to see whether the myocardial dysfunction was transient or persistent even after the stabilization of the patient. As far as it could be reviewed, no study relating BNP levels in pediatric asthma patients could be found in literature.

Echocardiographic changes in bronchial asthma regarding RT ventricular and Ltventricular function will be assessed According to some studies right ventricular (RV) systolic and diastolic dysfunction were detected, even in mild cases, by echocardiography. On the other hand, left ventricular (LV) dysfunction usually presents itself in severe asthmatic cases which may be reversible in acute conditions (5).

Some studies showed that there were no differences in echocardiographic findings regarding the ventricular function with the exception of RV wall thickness (6).

Asthma affects ventricular contractility in children. Although cardiac systolic function was found to be impaired in asthmatic patients, contrary to the literature diastolic dysfunction didn't observed in these patients even by tissue Doppler imaging, may be due to using inhaled corticosteroid(7). This was one of the most comprehensive studies among asthmatic patients. Further studies with larger sample sizes or without using corticosteroid treatment war ranted to better elucidate the cardiac function.

ELIGIBILITY:
Inclusion Criteria:

* all pediatric cases between the age of 5 -15years with acute severe bronchial asthma who were admitted in pediatric emergency care unit

Exclusion Criteria:

* Children with congenital or acquired heart diseases
* Foreign body aspiration .
* Chest infections
* Tuberculosis or pneumonia

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children aged from 5 years to 15 years diagnosed as bronchial asthma
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
to identify the relation between asthmatic children and cardiac function | Baseline
  relation between asthma and cardiac function
to identify the relation between asthmatic children and myocardial dysfunction | Baseline
  relation between asthma and myocardial dysfunction

OTHER OUTCOMES:
to identify the relation between asthmatic children and child weight | Baseline
  relation between asthma outcome and patient wieght

REFERENCES:
- [Background] Rodriguez-Roisin R, Ballester E, Roca J, Torres A, Wagner PD. Mechanisms of hypoxemia in patients with status asthmaticus requiring mechanical ventilation. Am Rev Respir Dis. 1989 Mar;139(3):732-9. doi: 10.1164/ajrccm/139.3.732. PMID 2923373
- [Background] Peng SM, Sun P, Zeng J, Deng XM. [Cardiac function of children with bronchial asthma]. Zhongguo Dang Dai Er Ke Za Zhi. 2006 Oct;8(5):388-90. Chinese. PMID 17052399
- [Background] Zeybek C, Yalcin Y, Erdem A, Polat TB, Aktuglu-Zeybek AC, Bayoglu V, Akdeniz C, Celebi A. Tissue Doppler echocardiographic assessment of cardiac function in children with bronchial asthma. Pediatr Int. 2007 Dec;49(6):911-7. doi: 10.1111/j.1442-200X.2007.02486.x. PMID 18045296
- [Background] Shedeed SA. Right ventricular function in children with bronchial asthma: a tissue Doppler echocardiographic study. Pediatr Cardiol. 2010 Oct;31(7):1008-15. doi: 10.1007/s00246-010-9753-2. Epub 2010 Aug 10. PMID 20697704
- [Background] Sears MR. Trends in the prevalence of asthma. Chest. 2014 Feb;145(2):219-225. doi: 10.1378/chest.13-2059. PMID 24493506